CLINICAL TRIAL: NCT05572112
Title: Post Market Clinical Follow-up Study on the Performance /Safety of Celsite® Venous Access Ports in Patients Who Need Repeated Venous Access
Brief Title: The Performance / Safety of the Celsite® Venous Access Ports
Acronym: CAP
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: B.Braun Médical - CoE Chasseneuil (Industry)
Responsible Party: Sponsor
Other Study IDs: AAG-0-H-2122
Record Dates: First submitted 2022-10-05; First posted 2022-10-07 (Actual); Last update posted 2022-10-07 (Actual); Status verified 2022-10

CONDITIONS: The Performance / Safety of the Celsite® Venous Access Ports

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Venous access port implantation — Venous access port implantation

SUMMARY:
The Celsite® Venous Access Ports System are intended to be used for repeated intravenous administration of, for example, chemotherapy, antibiotic and antiviral drugs, total parenteral nutrition, blood sampling or transfusion.

The objective is to assess the device's safety to deliver medication over the time in regard to the rate of adverse events related to the Celsite® access ports written in the IFU.

ELIGIBILITY:
Inclusion Criteria:

* Patient is at least 18 years old
* Provision of voluntary consent to participate in the study, following a full explanation of the nature and purpose of the study, by signing the informed consent form approved by the Ethics Committee (EC) prior to all evaluations.
* Patient for whom the access port placement has already been determined as the best treatment option within the regular planning of the patient's treatment in accordance with the IFU.
* Patients who are mentally and linguistically able to understand the aim of the study and to show sufficient compliance in the following study protocol

Exclusion Criteria:

* Patient for whom the technical and/ or clinical characteristics of the access port placement or use is outside the scope of the IFU.
* Patient not followed-up in the center where the access port is implanted.
* Pregnancy
* Patient < 18 years of age

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patient is at least 18 years old
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2022-10-15 (Estimated); Primary Completion 2023-01-30 (Estimated); Study Completion 2025-01-30 (Estimated)

PRIMARY OUTCOMES:
To assess the device's safety | 2 years
  The primary variable is the incidence/frequency of all adverse reactions/complications (intraoperative, postoperative, late etc.) which occurred during the study. Focus will be done on all adverse reactions/complications (intraoperative, postoperative, late etc.) related to the Celsite® access ports written in the IFU in comparison with the published data.

IPD SHARING:
Plan to Share IPD: No